CLINICAL TRIAL: NCT02349971
Title: Safety and Feasibility of MR-Guided High Intensity Focused Ultrasound (MR-HIFU) Ablation of Osteoid Osteoma in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Karun Sharma MD, MD, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU OO
Record Dates: First submitted 2015-01-15; First posted 2015-01-29 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Osteoid Osteoma
MeSH Terms: conditions — Osteoma, Osteoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Experimental): Patients will undergo a one-time procedure of MR-HIFU ablation of OO under sedation or anesthesia. Patients will be monitored for disease status and adverse events for at least 12 months following procedure.
  Interventions: Device: MR-HIFU

INTERVENTIONS:
Device: MR-HIFU — Magnetic Resonance guided High Intensity Focused Ultrasound (MR-HIFU) provides precise and controlled delivery of focused ultrasound energy inside a lesion using an external applicator, without the need for a scalpel or needle

SUMMARY:
This study looks to examine the feasibility and efficacy of using MR-HIFU to ablate Osteoid Osteoma lesions in children and young adults.

DETAILED DESCRIPTION:
Osteoid Osteoma (OO) is a benign, but painful, bone tumor commonly occurring in children and young adults. Common treatment options are surgical excision or, more recently, CT-guided radiofrequency ablation (RFA). RFA is less invasive, but it still requires drilling from the skin through muscle and soft tissue into bone. It also exposes the patient and operator to ionizing radiation.

Magnetic Resonance guided High Intensity Focused Ultrasound (MR-HIFU) provides precise and controlled delivery of focused ultrasound energy inside a lesion using an external applicator, without the need for a scalpel or needle. MR-HIFU has been successfully used to treat painful bone metastases in adult clinical trials and one recent report suggests that it can also be used to treat OO.

MR-HIFU ablation of OO may provide a better alternative to surgical resection or RFA as it is completely non-invasive and does not require ionizing radiation. These two qualities of MR-HIFU are especially beneficial in growing children and young adults. Furthermore, MR-HIFU OO ablation is quick, with expected total procedure time of less than two hours. Such short treatments offer additional safety benefits from reduced anesthesia / sedation requirement compared to surgery and RFA

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * All patients with a clinical suspicion of OO based on presence of typical symptoms of localized nocturnal pain that is relieved by NSAIDs and unrelated to trauma or activity.
  * Typical imaging findings on CT and/or MRI. Plain radiographs and bone scans may be obtained by referring physicians and are helpful for confirming the clinical diagnosis but cannot be substituted for a CT or MRI.
  * Non-contrast enhanced or contrast enhanced CT studies are acceptable.
  * Contrast enhanced MRI studies should be performed.
  * Tissue biopsy is not required
* Tumor location:

  * Target lesions can be located in any peripheral bone with acoustic accessibility.
  * Target lesions may be intracortical or juxtacortical in location.
  * Target lesions must be reachable within the normal safety margins of HIFU as specified in the instructions for use.
* Prior therapy:

  ●Patients with prior unsuccessful surgical resection or RFA are eligible for enrollment.
* Laboratory :

  * Hemoglobin > 9 g/dL
  * Platelet count ≥75,000/µL (may receive transfusions)
  * Normal PT, PTT and INR < 1.5 x ULN (including patients on prophylactic anticoagulation)
  * Renal function: Age-adjusted normal serum creatinine (table in protocol) OR a creatinine clearance ≥60 mL/min/1.73 m2 for safe contrast administration
* Adequate pulmonary function: Defined as no dyspnea at rest, and a pulse oximetry >94% on room air if there is clinical indication for determination.

Exclusion Criteria:

* Clinically significant unrelated systemic illness, such as serious infections, hepatic, renal or other organ dysfunction, which in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate the general anesthetic required for the procedure.
* Implant or prosthesis or scar tissue within the path of the HIFU beam.
* Target <1 cm from nerve plexus, spinal canal, bladder, bowel
* Target <1 cm of the growth plate (physis)
* Lesion in the skull or vertebral body
* Inability to undergo MRI and/or contraindication for MRI
* Inability to tolerate stationary position during HIFU
* Patients currently receiving any investigational agents.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-03 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility measured by the number of patients who are able to be treated with MR HIFU and do not experience significant treatment related adverse events. | 12 months
  Safety and feasibility will be measured by the number of patients who are able to be treated with MR HIFU and do not experience significant treatment related adverse events.

SECONDARY OUTCOMES:
Response | 12 months
  Provide an assessment of MR-HIFU ablation of OO in children by the number of patients who experience a measurable clinical and imaging response.

CONTACTS AND LOCATIONS:
Overall Officials: Karun Sharma, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Sharma KV, Yarmolenko PS, Celik H, Eranki A, Partanen A, Smitthimedhin A, Kim A, Oetgen M, Santos D, Patel J, Kim P. Comparison of Noninvasive High-Intensity Focused Ultrasound with Radiofrequency Ablation of Osteoid Osteoma. J Pediatr. 2017 Nov;190:222-228.e1. doi: 10.1016/j.jpeds.2017.06.046. Epub 2017 Aug 17. PMID 28823554